CLINICAL TRIAL: NCT04682834
Title: Expanded Access for the Use of Sulopenem Etzadroxil/Probenecid for the Treatment of Patients With Complicated Urinary Tract Infection Due to Quinolone-nonsusceptible Uropathogens
Brief Title: Expanded Access Use of Sulopenem Etzadroxil/Probenecid for Complicated Urinary Tract Infection
Status: No longer available | Type: Expanded Access
Sponsor: Iterum Therapeutics, International Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: IT001-307
Record Dates: First submitted 2020-12-18; First posted 2020-12-24 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Complicated Urinary Tract Infection; Acute Pyelonephritis
MeSH Terms: interventions — Probenecid

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Sulopenem Etzadroxil/Probenecid — Individual Patients
  Other Names: Individual Patients

SUMMARY:
Sulopenem etzadroxil/probenecid is available to clinicians through an Expanded Access Program for the treatment of complicated urinary tract infections due to quinolone nonsusceptible uropathogens after an initial course of effective intravenous therapy. The investigational product may be requested by sending an email to the Sponsor (EAProgram@iterumtx.com), as listed on the Reagan Udall EAP Navigator website (https://navigator.reaganudall.org/company-directory/i).

DETAILED DESCRIPTION:
This Expanded Access Program will allow clinicians to use sulopenem etzadroxil/probenecid for the treatment of patients with serious or immediately life-threatening complicated urinary tract infection due to quinolone-nonsusceptible uropathogens where there are no satisfactory oral alternatives to use as step-down therapy after receiving an initial course of effective intravenous therapy. The recommended dose of sulopenem etzadroxil/probenecid 500 mg/ 500 mg is one bilayer tablet orally twice daily, taken with food whenever possible. No dose adjustment is required for patients with renal impairment. Duration of therapy will be at the discretion of the prescribing clinician, depending on the type of infection being treated and the response to therapy, and is expected to be less than ten days total.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age with complicated urinary tract infection due to a quinolone-nonsusceptible uropathogen
2. Patient or the patient's legally acceptable representative able to provide a signed written informed consent prior to any study-specific procedures.
3. Clinically documented pyelonephritis or complicated urinary tract infection for which at least one dose of effective intravenous antibiotics has been received.

Exclusion Criteria:

1. Patients who require concomitant administration of valproic acid
2. Patients with known hypersensitivity to any component of this product or to other drugs in the same class or in patients who have demonstrated anaphylactic reactions to beta-lactam antibacterial drugs or probenecid.
3. Patients with known uric acid kidney stones
4. Patients requiring concomitant use of ketorolac tromethamine or ketoprofen

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult